CLINICAL TRIAL: NCT07108881
Title: Ultrasound Guided Fluid Loading Before Spinal Anesthesia for Cesarean Section in Hypovolemic Parturient: Double-Blind Randomized Controlled Trial
Brief Title: Ultrasound Guided Fluid Loading Before Spinal Anesthesia
Acronym: EHCOPRESPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, principal inverstigator, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 0123
Record Dates: First submitted 2025-07-29; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section Complications; Spinal Anesthesia; Hypotension; Hypovolemia; Sympathetic Blockade; Fluid Loading
MeSH Terms: conditions — Hypotension; Hypovolemia

STUDY DESIGN:
Intervention Model Description: hypovolemic participant were chosen among all pauturient scheduled for cesarean section. hypovolemia was detected using VTI variation mesurment in spine position with passive legs raising then they were randomized into two groups group C: had an ultrasound guided preloading with 1 to 4 fluid challenges of 250 ml of cristalloids each group T: received the standard care, ie: critalloids co-loading with recsue ephedrine doses if needed
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: participant was blinded outcome assessors performed ultrasound to assess volemia but later were not aware of randomization care givers did know about randomization in order to give treatement according to the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group C (Active Comparator): hypovolemic parturient receiving cardiac -ultrasound -VTI guided cristalloid preloading with 1 to 4 fluid challenges of 250 ml each until they reach a normal volemic state before receiving spinal anesthesia
  Interventions: Drug: C
- groupT (Placebo Comparator): hypovolemic parturient reiving the standard care ie; they dont receive any preloading but coloading with critalloids with rescue boluses of ephedrine if hypotension happens
  Interventions: Drug: T

INTERVENTIONS:
Drug: C — isotonic saline solution infusion (fluid preloading) to achieve correction of hypovolemia before spinal anesthesia using cardiac ultrasoud guidance by measurment of VTI variation after a 250ml saline solution loading, with a maximum of 4 challenges, until hypovolemia complete correction
  Other Names: isotonic saline solution preloading
  Arms: group C
Drug: T — isotonic saline solution coloading after spinal anesthesia associated with recsue boluses of Ephedrine would be the "standard of care" in this arm. No correction of hypovolemia is done before spinal anesthesia. parturients receive a cristalloid coloading with saline isotonic solution with rescue boluses of ephedrine if hypotesion happens after spinal anesthesia
  Other Names: isotonic saline solution coloading with ephedrine boluses
  Arms: groupT

SUMMARY:
Perioperative hypotension is a common complication of spinal anesthesia during cesarean sections.

The aim of this study was to evaluate the effectiveness of echoguided correction of hypovolemia through crystalloid preloading on the incidence of arterial hypotension during scheduled cesarean sections under spinal anesthesia.

It was a double-blind, randomized controlled trial study conducted on hypovolemic parturients, scheduled for cesarean section. investigators compared ultrasound guided correction of hypovolemia to a standard care protocol without preloading.

Hypovolemia was defined as a ≥12% increase in the variation of the velocity-time integral of subaortic blood flow during a passive leg raising test.

Preloading was guided by the variation of the velocity-time integral of subaortic blood flow during volume expansion tests.

DETAILED DESCRIPTION:
In the literature, numerous studies have compared the different pre-filling and co-filling protocols with different solutes. The majority of them conclude that co-filling is superior to pre-filling when the same type of solute is used. Pre-filling with crystalloids was then abandoned in favor of co-filling with crystalloids It is essential to remember that several invasive or non-invasive means of hemodynamic monitoring have previously been validated in pregnant women The use of invasive tools for assessing blood volume, particularly arterial and central venous catheters, is limited given the brevity of obstetric procedures, the risk of morbidity in awake patients and their high costs. Although non-invasive methods are preferable, some remain imperfect, notably carotid Doppler and bioimpedance devices Transthoracic echocardiography stands out as a particularly reliable and relevant non-invasive tool for assessing cardiac output and blood volume in parturients It allows analysis of the variation of the subaortic velocity time integral (∆ ITV s-a) during the passive leg raise test (LET). It is the only dynamic preload parameter validated in patients during spontaneous ventilation, thus allowing assessment of blood volume.

After reviewing the literature, the investigators found no studies about, exclusively hypovolemic patients, the effect of combining pre-filling with co-filling with crystalloids, monitored by echocardiographic preload-dependence indices, on the incidence of arterial hypotension during elective cesarean sections performed under spinal anesthesia.

In this study, monitoring was performed by transthoracic echocardiography, based on the variation in subaortic TVI following the passive leg raise test and vascular fluid tests.

The objective of this prospective randomized study was to evaluate the efficacy of ultrasound-guided correction of hypovolemia by pre-filling with crystalloids on the incidence of arterial hypotension during elective cesarean sections performed under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

ASA II score, singleton pregnancy cesarean section

Exclusion Criteria:

Spinal anesthesia failure general anesthesia postpartum hemorhage saline solution volume > 1000 ml for preloading echocardiography: difficulties Poor echogenicity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females sheduled for cesarean delivery
Enrollment: 116 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
incidence of post-spinal anesthesia arterial hypotension during surgery | 60 minutes
  The incidence of intraoperative post-spinal hypotension Defined by a drop in blood pressure (BP) of more than 20% of its reference value, or a blood pressure (BP) < 100 mmHg

SECONDARY OUTCOMES:
Time to onset of the first episode of arterial hypotension (min) | 60 minutes
  hypotension is Defined by a drop in SBP of more than 20% of its reference value, or a SBP < 100mmHg
Duration of hypotensive episode (min) | 60 minutes
  the duration of hypotension from the onset of the first episode until reaching normal ranges again
Depth of hypotension (% fall from baseline value) | 60 minutes
  hypotension is Defined by a drop in SBP of more than 20% of its baseline value, or a SBP < 100mmHg
Variation in intraoperative cardiac output (% drop from baseline) | 60 minutes
  cardiac output is expected to rise of fall from its baseline and is caculated in percenttages of variation from its baseline
Consumption of per-op vasopressors (mg of ephedrine) | 60 minutes
  total dose of ephedrine given in case of hypotension
Volume of cristalloids and colloids infused (ml) | 60 minutes
  total volume of critalloids given either when preloading bfeore spinal anesthesia or while coloading after spinal anesthesia
Incidence of maternal bradycardia (%) - | 60 minutes
  (Heart Rate < 50 bpm)
Incidence of intraoperative nausea and vomiting (%) | 60 minutess
  nausea and vomiting usually at the moments of severe hypotension
Fetal pH at the umbilical cord at birth. | 30 minutes
  right after delivery
Newborn APGAR score at the first and fifth minute | 30 minutes
  at birth

CONTACTS AND LOCATIONS:
Locations (1):
- Tunis maternity and neonatology center, minisetry of public health, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No